CLINICAL TRIAL: NCT04983199
Title: Patient Reported Outcomes/Metrics Program Trial - Palliative Radiation
Brief Title: Patient Reported Outcomes/Metrics Program Trial
Acronym: PROMPT
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 21-5322
Record Dates: First submitted 2021-07-08; First posted 2021-07-30 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Cancer; Palliative
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Hexoskin Medical System — Hexoskin is a smart shirt that can detect heart rates, lung function and physical activity of patients before and after radiotherapy.
  Other Names: Hexoskin Smart Shirt

SUMMARY:
This is an observational study to investigate if it is feasible to recruit 100 patients receiving radiotherapy (RT) to metastatic disease to wear Hexoskin and if Hexoskin will facilitate the monitoring, detection and early treatment of RT-related side effects.

DETAILED DESCRIPTION:
Radiotherapy is an important adjunct in the interdisciplinary care of the palliative patient population, providing the potential for improved quality of life and symptom control, often translating into improved well-being, function and mobility. Changes in pain and QOL are frequently measured subjectively using patient-reported questionnaires. Objective measures such as respiratory rate, pulse rate, activity level and sleep duration and quality, may complement the currently available tools. Such tools may lead to better evaluation of the effects of palliative RT with real-time detection of potential complications and toxicity and the acute need for analgesic adjustments that can result from successful palliative RT.

ELIGIBILITY:
Inclusion Criteria:

* Planned to receive palliative radiotherapy for pain
* Known cancer diagnosis
* Able to wear Hexoskin Medical Shirt
* Ability to use and populate the mobile app (Zamplo) with or without assistance
* ECOG: 0-3
* Willing to provide a list of analgesic (pain relief) medication
* Willing to complete questionnaires
* Life expectancy of at least 3 months

Exclusion Criteria:

* Receiving whole brain radiotherapy
* Major cognitive or psychiatric impairments
* Pregnant women
* Allergies to: polyester, synthetic fibers
* Patients with pacemakers or implantable cardioverter-defibrillator (ICD)
* Patients on a Holter Monitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients planned for palliative radiotherapy to metastatic disease.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Rate of patient accrual | Over 12 months
  Feasibility of accruing 100 patients to the study
Frequency of radiotherapy related adverse events | Baseline to 12 months
  Frequency of grade 2 or above radiotherapy related adverse events with extended monitoring.

SECONDARY OUTCOMES:
Quality Adjusted Life Years (QALY) | Baseline to 12 months
  Perform economic and health technology assessment using EuroQol-5 Dimension-5 Level (EQ-5D-5L) health questionnaire. (100 is the best health a patient can imagine while 0 is the worst health a patient can imgaine.)
Health Related Quality of Life (QOL) | Baseline to 12 months
  Perform Health Related Quality of Life using EORTC QLQ-C30 and rate electronic survey completion.
Number of Trial Refusals | Baseline to 12 months
  Evaluate reasons for trial refusal
Complete follow-ups | Baseline to 12 months
  Rate of completed follow-ups
Patient experience and satisfaction | Baseline to 12 months
  Measure patient experience and satisfaction using mobile app (Zamplo) and Hexoskin
Patient Adherence | Baseline to 12 months
  Patient adherence to using the Hexoskin Medical System
Hexoskin data collection rates | Baseline to 12 months
  Feasibility of data collection using the Hexoskin Medical System
Quality of Life (QOL) survey completion | Baseline to 12 months
  Rate of Quality of Life (QOL) survey completion on mobile app (Zamplo)
Overall survival of participants | Baseline to 12 months
  Overall survival time is calculated from study enrollment to date of death or last follow-up
Characterize adverse event profile | Baseline to 12 months
  Characterize adverse event profile of various radiotherapy regimens given for metastases

CONTACTS AND LOCATIONS:
Overall Officials: Philip Wong, Principal Investigator — The Princess Margaret Cancer Foundation
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Othman H, Hannon B, Liu ZA, Raman S, Sexton E, Kasper C, Auger H, Tsai CJ, Barry A, Wong P. Patient Reported Outcomes/Metrics Program Trial (PROMPT)-palliative radiation: protocol of a prospective observational feasibility study. Ann Palliat Med. 2025 Nov;14(6):570-578. doi: 10.21037/apm-25-19. PMID 41360655